CLINICAL TRIAL: NCT00761475
Title: Primary Mesh Closure of Abdominal Midline Wounds; a Prospective Randomized Multicenter Trial
Brief Title: Primary Mesh Closure of Abdominal Midline Wounds
Acronym: PRIMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Baxter Healthcare Corporation (Industry); Aesculap AG (Industry)
Responsible Party: Principal Investigator, Hasan Eker, Prof. Dr. J.F. Lange, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRIMA TRIAL
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Incisional Hernia Occurence
Keywords: incisional hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): primary closure of the midline
  Interventions: Procedure: primary closure
- 2 (Active Comparator): onlay mesh supported closure
  Interventions: Procedure: mesh supported closure
- 3 (Active Comparator): sublay mesh supported closure
  Interventions: Procedure: mesh supported closure

INTERVENTIONS:
Procedure: mesh supported closure — onlay mesh supported closure midline laparotomy
  Arms: 2
Procedure: primary closure — primary closure of the midline
  Arms: 1
Procedure: mesh supported closure — sublay mesh supported closure midline laparotomy
  Arms: 3

SUMMARY:
Incisional hernia is the most frequently seen long term complication in surgery causing much morbidity and even mortality in patients. Despite studies on the optimal closing technique for laparotomies, the risk for incisional hernia after midline incision remains about 5-20 %. Major risk factors for incisional hernia after a laparotomy, like obesity, steroid use, malnutrition, smoking and connective tissue disorders, are known. Despite this knowledge, there has not yet been developed a sufficient method for prevention. One specific group of high risk patients are patients with an abdominal aortic aneurysm (AAA). The relationship between aortic aneurysm and other abdominal wall hernias, like inguinal hernias, has been reported. Retrospective and prospective studies have shown an average risk for incisional hernia after AAA repair of 31.6 %. Another high risk group is the group of obese patients. Patients with a BMI of more than 27 have a high risk of developing an incisional hernia after midline incision with an incidence of 22% after 12 months. Considering only 50 % of incisional hernia will be clinically evident in the first 12 months, the total incidence will be above 30%. This high risk group of patients with obesitas and aneurysmatic disease can benefit most from prevention. Some small studies have been performed to evaluate the usefulness and safety of primary laparotomy wound closure with the aid of prosthetic mesh. These studies show a very low risk for incisional hernias and a low infection rate, even when used in contaminated wounds such as colostomal surgery. However, there has not been performed an adequate randomized controlled trial to study the prevention of incisional hernias. Our hypothesis is that incisional hernia prevention with use of prosthetic mesh after laparotomy is effective in patients with aortic aneurysm and in obese patients with a BMI of more than 27.

ELIGIBILITY:
Inclusion Criteria:

* Every elective midline laparotomy for patients with Abdominal Aortic Aneurysm and patients with a BMI of more than 27.
* Signed informed consent

Exclusion Criteria:

* Age < 18 years
* Emergency procedure
* Inclusion in other trials
* Aortic reconstruction for obstructive disease
* Life expectancy less than 24 months
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
incisional hernia occurence | 2 years

SECONDARY OUTCOMES:
complications | 1 month
post-operative pain | 1 month
quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: J.F. Lange, Professor, Principal Investigator — Erasmus Medical Center
Locations (12):
- Wilhelminenspital, Vienna, Austria
- Germany (4):
  - Berlin-Charite Universitatsklinikum, Berlin
  - Hamburg-Eppefdorf Universitatsklinikum, Hamburg
  - Heidelberg University Medical Center, Heidelberg
  - Munchen University Medical Center, München
- Netherlands (7):
  - Erasmus Medical Center, Rotterdam, South Holland
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Scheper Ziekenhuis, Emmen
  - Maasstad Ziekenhuis, Rotterdam
  - Sint Franciscus Gasthuis, Rotterdam
  - Maxima Medisch Centrum, Veldhoven
  - Isala klinieken, Zwolle

REFERENCES:
- [Derived] Van den Dop LM, Sneiders D, Yurtkap Y, Werba A, van Klaveren D, Pierik REGJM, Reim D, Timmermans L, Fortelny RH, Mihaljevic AL, Kleinrensink GJ, Tanis PJ, Lange JF, Jeekel J; PRIMA Trialist Group. Prevention of incisional hernia with prophylactic onlay and sublay mesh reinforcement vs. primary suture only in midline laparotomies (PRIMA): long-term outcomes of a multicentre, double-blind, randomised controlled trial. Lancet Reg Health Eur. 2023 Nov 22;36:100787. doi: 10.1016/j.lanepe.2023.100787. eCollection 2024 Jan. PMID 38188275
- [Derived] Jairam AP, Timmermans L, Eker HH, Pierik REGJM, van Klaveren D, Steyerberg EW, Timman R, van der Ham AC, Dawson I, Charbon JA, Schuhmacher C, Mihaljevic A, Izbicki JR, Fikatas P, Knebel P, Fortelny RH, Kleinrensink GJ, Lange JF, Jeekel HJ; PRIMA Trialist Group. Prevention of incisional hernia with prophylactic onlay and sublay mesh reinforcement versus primary suture only in midline laparotomies (PRIMA): 2-year follow-up of a multicentre, double-blind, randomised controlled trial. Lancet. 2017 Aug 5;390(10094):567-576. doi: 10.1016/S0140-6736(17)31332-6. Epub 2017 Jun 20. PMID 28641875
- [Derived] Timmermans L, Eker HH, Steyerberg EW, Jairam A, de Jong D, Pierik EG, Lases SS, van der Ham AC, Dawson I, Charbon J, Schuhmacher C, Izbicki JR, Neuhaus P, Knebel P, Fortelny R, Kleinrensink GJ, Jeekel J, Lange JF. Short-term results of a randomized controlled trial comparing primary suture with primary glued mesh augmentation to prevent incisional hernia. Ann Surg. 2015 Feb;261(2):276-81. doi: 10.1097/SLA.0000000000000798. PMID 24983993
- [Derived] Nieuwenhuizen J, Eker HH, Timmermans L, Hop WC, Kleinrensink GJ, Jeekel J, Lange JF; PRIMA Trialist Group. A double blind randomized controlled trial comparing primary suture closure with mesh augmented closure to reduce incisional hernia incidence. BMC Surg. 2013 Oct 28;13:48. doi: 10.1186/1471-2482-13-48. PMID 24499111